CLINICAL TRIAL: NCT00915044
Title: Characterization of Interactions Between Immune Cells of Intestinal Mucosa or Peripheral Blood With the Extracellular Matrix in IBD
Brief Title: Interactions Between Immune Cells of Intestinal Mucosa or Peripheral Blood With the Extracellular Matrix in Inflammatory Bowel Disease (IBD)
Acronym: IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Iris Dotan, Dep. of Gastroenterology, Tel Aviv medical center
Other Study IDs: TASMC-07-ID-153-CTIL; 153-07
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 15 ml peripheral blood will be obtained from all participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBD patients: Approximately 40 patients (adults and children) suffering from IBD will be enrolled.
- Controls: Approximately 100 healthy controls

SUMMARY:
The purpose of this study is to examine the effects of different environmental factors on immune cells in patients with IBD.

DETAILED DESCRIPTION:
Background: Inflammatory bowel diseases, comprised of Crohn's Disease (CD) and ulcerative colitis (UC) are idiopathic disorders caused due to immunological, genetic, and environmental factors. These disorders are fairly common (in the US, there are 11 cases of CD and 7 cases of UC for every 100,000 people). The frequency of IBD, especially CD, are constantly rising (1). Clinical symptoms include diarrhea, rectal bleeding, abdominal pain, intestinal obstructions, and fistulas in CD. There are also systemic manifestations such as fever, weight loss, and anemia. The current hypothesis of IBD pathogenesis is an aberrant, ongoing, uncontrolled inflammatory response of the intestine, caused by commensal microbiota. The inflammatory response in IBD is mediated by T cells; in CD the pathologic lymphocytes are CD4 cells of Th1 type, while UC is considered an atypical Th2 response (2). CD4 T cells have a major role in initiation of inflammatory response in the gut, as well as a role in propagation and control of the inflammation.

Chemokines are low-molecular weight cytokines with chemoattractant capacity, and have a role in many inflammatory disorders. The chemokine CXCL12 is considered to be constitutively expressed (3). Our group found increased expression of CXCL12 in IBD (REF?). This finding suggests that CXCL12 might have a role in inflammatory processes of the gut.

Understanding phenotypical and functional differences of lymphocytes in mucosal homeostasis and IBD, elucidation of factors causing these differences, and recognition of causes for increased CXCL12 expression, will enable to increase knowledge of IBD; as well as lead to development of future therapeutic interventions in IBD.

Research Goals: To examine the effects of different environmental factors (cytokines, chemokines, extracellular matrix moieties) on immune cells from peripheral or intestinal source (in homeostasis or IBD) in terms of phenotypical and functional parameters.

Methods: 15 ml peripheral blood will be obtained from all participants. T lymphocytes will be isolated for the different experiments. Methods will include: Migration towards chemokines using the Transwell assay, proliferation will be assessed by either BrdU or thymidine incorporation, cytokine secretion will be determined using ELISA, phenotypical characterization will be done using flow cytometry and adhesion assays.

Ages: Adults and children aged 10-80. Research group: Approximately 40 patients (adults and children) suffering from IBD will be enrolled.

Control group: Approximately 100 controls will be enrolled in the research.

ELIGIBILITY:
Inclusion Criteria:

* IBD

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children aged 10-80. Research group: Approximately 40 patients (adults and children) suffering from IBD will be enrolled.
  Control group: Approximately 100 controls will be enrolled in the research.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Migration towards chemokines,proliferation, cytokine secretion, phenotypical characterization. | Once, when joining the study

CONTACTS AND LOCATIONS:
Overall Officials: Iris Dotan, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Dep. of Gastroenterology, Tel Aviv medical center, Tel Aviv, Israel